CLINICAL TRIAL: NCT06899165
Title: Processing Intergenerational Trauma With Psilocybin-Assisted Therapy
Brief Title: Psilocybin-Assisted Therapy for Intergenerational Trauma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rachel Yehuda (Other)
Responsible Party: Sponsor-Investigator, Rachel Yehuda, Director of the Parsons Research Center for Psychedelic Healing, Professor of Psychiatry at Mount Sinai, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-01320
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Psychological Stress; Depression; Anxiety
Keywords: psilocybin; psilocybin-assisted therapy; intergenerational trauma; psychedelic; stress; genocide
MeSH Terms: conditions — Stress, Psychological; Depression; Anxiety Disorders; Historical Trauma | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psilocybin-Assisted Therapy (Experimental): Offspring of genocide survivors with mood and anxiety disorders will undergo weekly therapy sessions and will be given 2 doses of psilocybin at least 3 weeks apart.
  Interventions: Drug: Psilocybin; Behavioral: Integration sessions

INTERVENTIONS:
Drug: Psilocybin — Psilocybin 25mg, capsules taken orally under the supervision of two trained study therapists
  Other Names: Psilocybin-Assisted Therapy
Behavioral: Integration sessions — weekly integration sessions (therapy) for 6 weeks

SUMMARY:
This is an open-label psilocybin-assisted therapy study that will examine the safety and tolerability of psilocybin-assisted therapy in the offspring of genocide survivors with mood and anxiety disorders.

The study will also investigate the efficacy of psilocybin-assisted therapy in reducing symptoms such as depression, anxiety and stress, as well as changes to the psychological effects of parental exposure to genocide, and changes to psychological resilience.

DETAILED DESCRIPTION:
This study is investigating whether Psilocybin-assisted therapy improves depression, anxiety and stress symptoms in the offspring (biological children) of genocide survivors. Intergenerational trauma is the concept that the effects of experiencing extreme stress can be perpetuated to future generations. A genocide here is defined by the extinction or threat of extinction of a racial, religious or ethnic group, by an oppressive regime. A genocide survivor here is defined by an individual who survived or escaped a genocide in their country of origin. Currently, there are no evidence-based treatments developed specifically for the syndrome associated with Intergenerational trauma. This study aims to assess the safety and tolerability of psilocybin-assisted therapy, and assess the efficacy of psilocybin-assisted therapy in reducing symptoms such as depression, anxiety and stress, as well as changes to the psychological effects of parental exposure to genocide, and changes to psychological resilience.

Participants will be asked to attend one or more screening visits to assess eligibility. If eligible, participants will be treated with two separate doses of the study medication, Psilocybin, 3-4 weeks apart. This is an open-label research study, meaning all participants will receive Psilocybin (25mg). Two trained clinical practitioners will work with participants across preparation, dosing, and integration processes. Participants will complete assessments throughout the study until their participation has ended. Safety measures are in place to check the overall health and well-being of participants

Participation will consist of:

* Screening Period (up to 4 weeks): Phone screen, informed consent, eligibility assessment.
* Tapering & Enrollment Period (variable): Enrollment, supervised medical tapering where necessary as discussed with the study doctor, biomarker collection and psychometric baseline assessments.
* Preparatory & Treatment Period (up to 14 weeks): Three preparatory sessions with study clinicians, assessments; two dosing days at least three weeks apart, three weekly integration sessions with study clinicians following each dose, a 72-hour check-in call after each dosing day, assessments.
* Follow-Up Period (up to 5 weeks): Follow-up one month after final integration session, assessments, clinical evaluation, biomarker collection

ELIGIBILITY:
Inclusion criteria:

* Age at least 18 years old at time of signing the informed consent
* Biological child of at least one parent who directly survived/escaped a genocide
* Meets diagnostic criteria for a depressive or anxiety disorder
* Capable of providing informed consent and complying with study procedures
* Currently using or agreeing to use adequate contraceptive methods.
* Fluent in speaking and reading English
* Able to swallow pills
* Agrees to have study visits recorded with audio and video
* Able to provide a contact person who can be reached by investigators in the event of the participant becoming unwell or unreachable
* Agrees to inform the investigators within 48 hours of any medical conditions and procedures
* Agrees to release of outside medical and psychiatric records
* Must not participate in any other interventional clinical trials for the duration of the study.
* Must commit to medication dosing, therapy, and all study procedures.

Exclusion Criteria:

* Not able to give adequate informed consent.
* Was directly exposed to or survived a genocide.
* Has a history of any medical condition, or any significant clinical finding on screening tests, that could make receiving psilocybin harmful.
* Has acute, severe or unstable medical illness.
* Has a history of stroke or Transient Ischemic Attack (TIA).
* Has a history of psychiatric hospitalization within the last 6 months.
* Current serious suicide risk.
* Unable or unwilling to safely taper off prohibited psychiatric medications.
* Abusing alcohol or other substances.
* Has used psychedelics within 3 months of enrollment.
* Are pregnant or nursing or able to become pregnant and are not practicing an effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2030-01-02 (Estimated)

PRIMARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS) | up to 23 weeks
  Suicide risk as determined by the Columbia-Suicide Severity Rating Scale (C-SSRS) - Full Scale: 0 - 6. Higher scores indicate increased risk of suicide.
Brief Psychiatric Rating Scale (BPRS-6) | up to 23 weeks
  Brief Psychiatric Rating Scale (BPRS-6) - Full Scale: 0 - 36. Higher scores indicate the number and severity of psychiatric symptoms.

SECONDARY OUTCOMES:
Change in Depression, Anxiety, and Stress Symptoms Scale (DASS-21) | Baseline (V0), Weeks Week 4-10 (V7), Week 6-15 (V11), Week 23(V12)
  Change in Depression, Anxiety, and Stress Symptoms Scale (DASS-21) score. Stress scale - Subscale: 0 - 42 Anxiety scale - Subscale: 0 - 42 Depression scale - Subscale: 0 - 42 Full scale: 0 - 126
  Higher scores indicate higher severity of symptomology.
Change in Parental PTSD Questionnaire (PPQ) | Baseline (V0) and Week 23 (V12)
  Change in Parental PTSD Questionnaire (PPQ) score. Full Scale: 11 - 55 Higher scores indicate more negatively affected by perception of parents' trauma
Change in Resilience Scale for Adults (RSA) | Baseline (V0) and at Week 23 (V12)
  Change in Resilience Scale for Adults (RSA) score. Full Scale: 33- 231 Higher scores indicate higher resilience

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Yehuda, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Parsons Research Center for Psychedelic Healing, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plans to at this time